CLINICAL TRIAL: NCT01230801
Title: A Phase 1/2 Open-label Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamic and Preliminary Efficacy of BMN 701 (GILT-tagged Recombinant Human GAA) in Patients With Late-onset Pompe Disease
Brief Title: Safety/Tolerability/Pharmacokinetic (PK)/Pharmacodynamics (PD) Study of BMN701 in Patients With Late-Onset Pompe Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POM-001; 2010-023561-22 (EudraCT Number)
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMN 701 (Experimental): IV infusion
  Interventions: Biological: BMN 701

INTERVENTIONS:
Biological: BMN 701 — GILT-tagged recombinant human GAA

SUMMARY:
A Phase 1/2, open-label, multicenter, multiple dose escalation study of BMN 701 administered by intravenous infusion every 2 weeks over a 24-week treatment period to patients with late-onset Pompe disease.

ELIGIBILITY:
Inclusion criteria:

* Patient has been diagnosed with Pompe Disease prior to or during the screening period based on 2 GAA gene mutations and either: endogenous GAA activity <75% of the lower limit of the normal adult range reported by the testing laboratory, as assessed in cultured skin fibroblasts -or- endogenous GAA activity <75% of the lower limit of the normal adult range reported by the testing laboratory, as assessed by dried blood spot or whole blood assay;
* Patient is male or female and 13 years of age or older at the time of enrollment in the study;
* Sexually active patients must be willing to use an acceptable method of contraception while participating in the study and for at least 4 months following the last dose of BMN 701;
* If patient is female and not considered to be of childbearing potential, she is at least 2 years post-menopausal or had tubal ligation at least 1 year prior to screening, or who have had total hysterectomy;
* If patient is female and of childbearing potential, she has negative urine pregnancy tests during the Screening Period and at the Baseline visit and be willing to have additional pregnancy tests during the study;
* Patient has ≥30% predicted upright FVC and either <80% predicted upright FVC, or >10% reduction in supine FVC compared to upright FVC during the Screening Period;
* Patient is naïve to Enzyme Replacement Therapy (ERT) with rhGAA;
* Patient must be able to ambulate at least 40 meters (131.2 feet) on the 6MWT conducted at the Screening visit (use of assistive devices such as walker, cane, or crutches, is permitted); and
* If subject was female, she was not lactating

Exclusion criteria:

* Patient has a history of diabetes or other disease known to cause hypoglycemia and is currently receiving, or might anticipate receiving, hypoglycemic agents during the course of the study;
* Patient has been on any immunosuppressive medication other than glucocorticosteroids within 1 year prior to enrollment into this study;
* Patient requires invasive ventilatory assistance at the time of enrollment into the study;
* Patient has received any investigational medication within 30 days prior to the first dose of study drug or is scheduled to receive any investigational drug other than BMN 701 during the course of the study;
* Patient has previously been admitted to the study;
* Patient is breastfeeding at screening or planning to become pregnant (self or partner) at any time during the study;
* Patient has a medical condition or extenuating circumstance that, in the opinion of the Investigator, might compromise the patient's ability to comply with the protocol requirements or compromise the patient's well being or safety;
* Patient has any condition that, in the view of the Investigator, places the patient at high risk of poor treatment compliance or of not completing the study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01-17 (Actual); Primary Completion 2013-03-06 (Actual); Study Completion 2013-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — BioMarin Pharmaceutical
Locations (10):
- United States (3):
  - Univ of California San Diego School of Medicine, La Jolla, California
  - University of Florida College of Medicine, Gainesville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
- Royal Adelaide Hospital, SA Pathology, Adelaide, Adelaide, SA, Australia
- France (2):
  - Hôpital de I´Archet- Centre Hospitalier Universitaire Nice, Nice
  - Hôpital Pitié-Salpêtrière, Paris
- Zentrum für Kinder- und Jugenmedizin, Mainz, Rhineland-Palatinate, Germany
- United Kingdom (3):
  - Old Queen Elizabeth Hospital, Department of Medicine, Birmingham
  - Royal Free Hospital, London
  - Salford Royal Hospital NHS Trust, Salford

RESULTS

PARTICIPANT FLOW:
Groups:
- BMN 701 5 mg/kg: BMN 701 5 mg/kg IV
- BMN 701 10 mg/kg: BMN 701 10 mg/kg IV
- BMN 701 20 mg/kg: BMN 701 20 mg/kg IV
Period: Overall Study
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Started | 3 | 3 | 16
Completed | 3 | 3 | 15
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 16 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 16 | 22
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (6.81) | 42.3 (12.90) | 50.1 (5.37) | 49.3 (7.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 6 | 8
  Male | 3 | 1 | 10 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 2 | 16 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 15 | 21
  Other | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 0 | 0 | 4 | 4
  France | 0 | 0 | 2 | 2
  Germany | 0 | 0 | 1 | 1
  United Kingdom | 0 | 0 | 6 | 6
  United States | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events as a Measure of Safety and Tolerability
Time Frame: 24 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 3 | 3 | 16
Participants | 3 | 3 | 15

2. Secondary Outcome: Change From Baseline in Six Minutes Walk Test
Description: Change from Baseline in Six Minutes Walk Test. The 6MWT measured the maximum distance the subject could walk on a flat, hard surface in a period of 6 minutes
Time Frame: Baseline up to 24 weeks
Population: ITT Population. As some patients did not attend or all tests were not completed at each visit, some time points had different numbers of patients analyzed. The total number of patients analyzed for each arm is listed as the maximum patients analyzed at any given time point.
Measure: Mean (Standard Deviation); unit: meter
Groups:
- Total: Total Results
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 16 | 22
meter
  Baseline | 334 (227.12) | 360 (51.4) | 354.5 (156.94) | 352.5 (151.05)
  Change from Baseline - Week 6: number analyzed (Participants) | 2 | 3 | 16 | 21
  Change from Baseline - Week 6 | -2.5 (23.33) | -30.3 (56.50) | 19.8 (35.11) | 10.5 (40.08)
  Change from Baseline - Week 12: number analyzed (Participants) | 3 | 3 | 15 | 21
  Change from Baseline - Week 12 | 31.2 (78.81) | -13.7 (8.04) | 11.1 (42.67) | 10.4 (45.32)
  Change from Baseline - Week 18: number analyzed (Participants) | 3 | 3 | 15 | 21
  Change from Baseline - Week 18 | 43.3 (89.44) | -79.0 (104.61) | 16.4 (55.09) | 6.6 (73.43)
  Change from Baseline - Week 24 | 36.0 (76.02) | -42.7 (12.57) | 22.3 (54.23) | 15.3 (56.97)

3. Other Pre Specified Outcome: Change From Baseline in Percent Predicted Upright Forced Vital Capacity
Description: Change from Baseline in Percent Predicted Upright Forced Vital Capacity. Changes in respiratory function were assessed by measurement of MEP, MIP and MVV; and percent predicted upright and supine FVC.
Time Frame: Baseline up to 24 week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of Predicted Upright FVC
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 16 | 22
percentage of Predicted Upright FVC
  Baseline | 69.3 (19.73) | 67.3 (26.58) | 58.1 (18.42) | 60.9 (19.21)
  Change from Baseline - Week 6: number analyzed (Participants) | 2 | 3 | 16 | 21
  Change from Baseline - Week 6 | 4.0 (4.24) | -2.0 (2.65) | 0.4 (3.3) | 0.4 (3.46)
  Change from Baseline - Week 12 | -2.6 (9.5) | -3.7 (2.89) | 1.6 (4.35) | 0.3 (5.25)
  Change from Baseline - Week 18: number analyzed (Participants) | 3 | 3 | 15 | 21
  Change from Baseline - Week 18 | 1.5 (4.09) | 0.3 (3.06) | 1.2 (4.49) | 1.1 (4.1)
  Change from Baseline - Week 24 | 1.0 (2.65) | -1.7 (3.06) | 1.2 (3.89) | 0.8 (3.65)

4. Other Pre Specified Outcome: Change From Baseline in Percent Predicted Supine Forced Vital Capacity
Description: Change from Baseline in Percent Predicted Supine Forced Vital Capacity. Changes in respiratory function were assessed by measurement of MEP, MIP and MVV; and percent predicted upright and supine FVC.
Time Frame: Baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of Predicted Supine FVC
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 16 | 22
percentage of Predicted Supine FVC
  Baseline: number analyzed (Participants) | 3 | 3 | 13 | 19
  Baseline | 36.7 (17.95) | 47.7 (32.58) | 46.3 (21.93) | 45 (22.1)
  Change from Baseline - Week 6: number analyzed (Participants) | 2 | 3 | 13 | 18
  Change from Baseline - Week 6 | 2.1 (1.2) | -1.3 (4.04) | -0.8 (4.86) | -0.6 (4.44)
  Change from Baseline - Week 12: number analyzed (Participants) | 3 | 3 | 12 | 18
  Change from Baseline - Week 12 | 0.3 (4.22) | -4.7 (2.89) | 3.3 (3.87) | 1.5 (4.7)
  Change from Baseline - Week 18: number analyzed (Participants) | 3 | 3 | 12 | 18
  Change from Baseline - Week 18 | 1.3 (1.53) | -1.3 (6.66) | 2.3 (3.14) | 1.5 (3.7)
  Change from Baseline - Week 24: number analyzed (Participants) | 3 | 3 | 13 | 19
  Change from Baseline - Week 24 | 2.0 (3.0) | -3.3 (5.51) | 1.1 (4.42) | 0.5 (4.53)

5. Other Pre Specified Outcome: Change From Baseline in Percent Predicted Upright Maximum Expiratory Pressure
Description: Change from Baseline in Percent Predicted Upright Maximum Expiratory Pressure. Changes in respiratory function were assessed by measurement of MEP, MIP and MVV; and percent predicted upright and supine FVC.
Time Frame: Baseline up to 24 weeks
Population: ITT Population. As some patients did not attend or all tests were not completed at each visit, some time points had different numbers of patients analyzed. The total number of patients analyzed for each arm is listed as the maximum patients analyzed at any given time point. No patient had baseline assessment in group of BMN 701 5 mg/kg.
Measure: Mean (Standard Deviation); unit: percentage of Predicted MEP
Groups:
- Total: Total IV
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg | Total
Number analyzed (Participants) | 0 | 3 | 16 | 22
percentage of Predicted MEP
  Baseline: number analyzed (Participants) | 0 | 3 | 16 | 19
  Baseline |  | 31.1 (6.64) | 36.3 (15.46) | 35.5 (14.42)
  Change from Baseline - Week 6: number analyzed (Participants) | 0 | 3 | 16 | 19
  Change from Baseline - Week 6 |  | 6.8 (4.06) | 3.2 (5.38) | 3.8 (5.27)
  Change from Baseline - Week 12: number analyzed (Participants) | 0 | 3 | 16 | 19
  Change from Baseline - Week 12 |  | 1.4 (4.53) | 2.2 (8.68) | 2.0 (8.07)
  Change from Baseline - Week 18: number analyzed (Participants) | 0 | 3 | 16 | 19
  Change from Baseline - Week 18 |  | 1.2 (2.06) | 6.9 (7.21) | 6.0 (6.94)
  Change from Baseline - Week 24: number analyzed (Participants) | 0 | 3 | 16 | 19
  Change from Baseline - Week 24 |  | 2.5 (10.4) | 5.2 (8.25) | 4.8 (8.36)

6. Other Pre Specified Outcome: Change From Baseline in Percent Predicted Upright Maximum Inspiratory Pressure
Description: Change from Baseline in Percent Predicted Upright Maximum Inspiratory Pressure. Changes in respiratory function were assessed by measurement of MEP, MIP and MVV; and percent predicted upright and supine FVC.
Time Frame: Baseline up to 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of Predicted MIP
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg | Total
Number analyzed (Participants) | 0 | 3 | 16 | 22
percentage of Predicted MIP
  Baseline: number analyzed (Participants) | 0 | 3 | 16 | 19
  Baseline |  | 39.5 (21.87) | 40.5 (25.01) | 40.3 (23.97)
  Change from baseline at week 6: number analyzed (Participants) | 0 | 3 | 16 | 19
  Change from baseline at week 6 |  | 1.7 (1.46) | 5.3 (9.8) | 4.7 (9.06)
  Change from baseline at week 12: number analyzed (Participants) | 0 | 3 | 16 | 19
  Change from baseline at week 12 |  | 3.4 (6.74) | 11.4 (10.92) | 10.1 (10.65)
  Change from baseline at week 18: number analyzed (Participants) | 0 | 3 | 15 | 18
  Change from baseline at week 18 |  | 2.9 (11.77) | 14.5 (14.48) | 12.6 (14.45)
  Change from baseline at week 24: number analyzed (Participants) | 0 | 3 | 16 | 19
  Change from baseline at week 24 |  | 0.7 (6.69) | 11.1 (8.31) | 9.5 (8.81)

7. Other Pre Specified Outcome: Change From Baseline in Upright Maximum Ventilatory Volume
Description: Change from Baseline in Upright Maximum Ventilatory Volume. Changes in respiratory function were assessed by measurement of MEP, MIP and MVV; and percent predicted upright and supine FVC.
Time Frame: Baseline up to 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg | Total
Number analyzed (Participants) | 0 | 3 | 16 | 22
L/min
  Baseline: number analyzed (Participants) | 0 | 3 | 16 | 19
  Baseline |  | 76 (41.04) | 67.6 (25.9) | 68.9 (27.5)
  Change from Baseline - Week 6: number analyzed (Participants) | 0 | 3 | 16 | 19
  Change from Baseline - Week 6 |  | -1.0 (0.35) | 1.5 (11.1) | 1.1 (10.18)
  Change from Baseline - Week 12: number analyzed (Participants) | 0 | 3 | 16 | 19
  Change from Baseline - Week 12 |  | -1.1 (2.73) | 3.8 (11.64) | 3.0 (10.82)
  Change from Baseline - Week 18: number analyzed (Participants) | 0 | 3 | 15 | 18
  Change from Baseline - Week 18 |  | -3.9 (2.86) | 4.7 (10.89) | 3.3 (10.46)
  Change from Baseline - Week 24: number analyzed (Participants) | 0 | 3 | 15 | 18
  Change from Baseline - Week 24 |  | -0.7 (9.1) | 2.3 (10.71) | 1.8 (10.28)

ADVERSE EVENTS:
Time Frame: 32 weeks (27 days of screening and baseline measurements + 24 weeks of treatment + 20 days of follow-up)
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg | Total
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/16 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 4/16 | 4/22
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 15/16 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 701 5 mg/kg (N=3) | BMN 701 10 mg/kg (N=3) | BMN 701 20 mg/kg (N=16) | Total (N=22)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 701 5 mg/kg (N=3) | BMN 701 10 mg/kg (N=3) | BMN 701 20 mg/kg (N=16) | Total (N=22)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 3 (4) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 4 (16) | 5 (18)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (5) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (15) | 8 (15)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (9) | 7 (11)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (6) | 1 (2) | 5 (6) | 7 (14)
Chills (General disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Infusion site discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tenderness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaccination site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0) | 2 (3) | 3 (5)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (4) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 3 (5) | 3 (4) | 7 (11)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Complement factor decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory rate increased (Investigations) | 0 (0) | 0 (0) | 1 (5) | 1 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 14 (41) | 14 (41)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 2 (3) | 4 (7)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 6 (9) | 7 (10)
Headache (Nervous system disorders) | 1 (2) | 2 (8) | 6 (27) | 9 (37)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 5 (10) | 6 (12)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (5) | 4 (5)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (4) | 2 (5)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (13) | 2 (14)
Flushing (Vascular disorders) | 1 (5) | 0 (0) | 1 (1) | 2 (6)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 3 (5) | 3 (5)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Poor venous access (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days